CLINICAL TRIAL: NCT01806415
Title: A Double Blind, Randomized, Single Dose, Placebo Controlled Study of the Pharmacokinetics and Side Effects of the mGlu5 Antagonist Fenobam in Adult Healthy Volunteers
Brief Title: Pharmacokinetics and Side Effects of the mGlu5 Antagonist Fenobam in Adult Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Principal Investigator, Laura Cavallone, Assistant Professor of Anesthesiology, Washington University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: Triple
Other Study IDs: 201304126
Record Dates: First submitted 2013-03-02; First posted 2013-03-07 (Estimated); Last update posted 2015-12-09 (Estimated); Status verified 2015-12

CONDITIONS: Healthy
Keywords: Fenobam,; Pharmacokinetics; side effects
MeSH Terms: interventions — fenobam; Lactose

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Fenobam 50 mg (Experimental): Treatment regimen 1: Fenobam [1-(3-chlorophenyl)-3-(1-methyl-4-oxo-2-imidazolidinylidine) urea hydrate], oral administration of one 50 mg gelatin capsule.
  Interventions: Drug: Fenobam
- Fenobam 100 mg (Experimental): Treatment regimen 2: Fenobam, oral administration of one 100 mg gelatin capsule.
  Interventions: Drug: Fenobam
- Fenobam 150 mg (Experimental): Treatment regimen 3: Fenobam, oral administration of one 150 mg gelatin capsule.
  Interventions: Drug: Fenobam
- Placebo arm (Placebo Comparator): Treatment regimen 4: Placebo (lactose), oral administration of one 150 mg gelatin capsule.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Fenobam — Oral administration of 50, 100, or 150mg of Fenobam or placebo (lactose)
  Other Names: N-(3-chlorophenyl)-N'-(4,5-dihydro-1-methyl-4-oxo-1H-imidazole-2-yl)urea
  Arms: Fenobam 100 mg; Fenobam 150 mg; Fenobam 50 mg
Drug: Placebo — Oral administration of placebo or lactose 150 mg
  Other Names: Lactose
  Arms: Placebo arm

SUMMARY:
This is a randomized, blinded, parallel group, placebo-controlled trial on 32 evaluable healthy male and non-pregnant female, 18-50 year old volunteers. The investigators goal is to observe the pharmacokinetics of fenobam after oral administration of 50, 100 or 150 mg in groups of healthy individuals and to compare the side effects and tolerability of a single dose of fenobam with placebo.

DETAILED DESCRIPTION:
Treatment regimen 1: Fenobam [1-(3-chlorophenyl)-3-(1-methyl-4-oxo-2-imidazolidinylidine) urea hydrate], oral administration of one 50 mg gelatin capsule.

Treatment regimen 2: Fenobam, oral administration of one 100 mg gelatin capsule.

Treatment regimen 3: Fenobam, oral administration of one 150 mg gelatin capsule.

Treatment regimen 4: Placebo (lactose), oral administration of one 150 mg gelatin capsule.

ELIGIBILITY:
Inclusion Criteria

1. 18-50 yr old
2. Good general health with no remarkable medical conditions (e.g liver, kidney, heart, or lung failure), BMI<33 and no known drug allergies.
3. Willing to comply with study guidelines as outlined in protocol
4. Willing to provide informed consent.

Exclusion Criteria

1. Medication use (prescription or non prescription medications, vitamins, herbals, dietary and mineral supplements and grapefruit products during or within 14 days prior to study participation; excludes contraceptives)
2. History of addiction to drugs or alcohol (prior or present addiction or treatment for addiction)
3. Pregnant or nursing female
4. Lactose intolerance
5. Smokers

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2013-05; Primary Completion 2014-03 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic data after oral administration of 50, 100 or 150 mg of fenobam in groups of healthy individuals. | 24 hours
  Blood samples will be drawn periodically before and after fenobam/placebo administration for approximately 10 hours (at approximately 30, 60, 120, 180, 240, 300, 360 and 600 minutes) and one more time the next day (day 2).

SECONDARY OUTCOMES:
Number of participants with adverse events as a measure of tolerability | 1 week
  Participants will be administered a questionnaire regarding side effects at the end of the study day, after administration of a single dose of 50 mg, 100 mg or 150 mg of fenobam, or 150 mg placebo. The questionnaire will be administered again the following day and one week after the study day. Side effects in the fenobam treatment groups will be compared to side effects in the placebo group.

CONTACTS AND LOCATIONS:
Overall Officials: Laura Cavallone, MD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School Of Medicine, St Louis, Missouri, United States